CLINICAL TRIAL: NCT05620667
Title: Effects of Citrus Reticulate Unripe Fruit Extraction on Body Weight and Body Fat in Human Trial.
Brief Title: Effects of Citrus Reticulate Unripe Fruit Extraction on Body Weight and Body Fat.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chung Shan Medical University (Other)
Collaborators: TCI Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Chin-Lin Hsu, Professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CS2-22066
Record Dates: First submitted 2022-11-10; First posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- placebo (Placebo Comparator): Placebo 25mL, without any ingredients of immature ponkan extract. Drink 25mL for once, and once a day.
  Interventions: Dietary Supplement: placebo
- immature ponkan (Citrus reticulate) extract (Experimental): Immature ponkan (Citrus reticulate) extract 25 mL, drink 25mL for once, and once a day.
  Interventions: Dietary Supplement: immature ponkan (Citrus reticulate) extract
- immature ponkan (Citrus reticulate) extract with time restricted feeding (Experimental): Immature ponkan (Citrus reticulate) extract 25 mL, drink 25mL for once, and once a day, adding time restricted feeding.
  Interventions: Dietary Supplement: immature ponkan (Citrus reticulate) extract; Behavioral: time restricted feeding

INTERVENTIONS:
Dietary Supplement: immature ponkan (Citrus reticulate) extract — Drink 25mL for once, and once a day.
  Arms: immature ponkan (Citrus reticulate) extract; immature ponkan (Citrus reticulate) extract with time restricted feeding
Dietary Supplement: placebo — Drink 25mL for once, and once a day.
  Arms: placebo
Behavioral: time restricted feeding — Controlling a shortened period of time for eating within 8 hour each day.
  Arms: immature ponkan (Citrus reticulate) extract with time restricted feeding

SUMMARY:
The aim of this study is to investigate the effects of immature ponkan (Citrus reticulate) extract on body weight and body fat in overweight and obese adults.

DETAILED DESCRIPTION:
This randomized, placebo-controlled clinical trial will be conduct for 8 weeks with three hundred adults. Subjects will be recruited and randomly assigned into three groups: (1) placebo, n = 100; (2) immature ponkan extract, n=100; (3) immature ponkan extract with time restricted feeding, n=100. During the 8 weeks intervention, the subjects should take 25mL liquid of placebo or immature ponkan extract a day (drink 25mL for once, and once a day). The two drinks are supplied in aluminum foil packages, and both the products taste the same. Subjects also should complete the assessment of anthropometric measurement, intestinal questionnaire , food record, feces and blood collection at week 0, 4 and week 8.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* aged 20-60 years old
* body mass index is greater than or equal to 24 kg/m2, or body fat more than 30%

Exclusion Criteria:

* Subjects diagnosed with cancer and on curative care.
* Subjects diagnosed with heart disease and on curative care.
* Subjects who use other drugs whose pharmacological effects may affect the experiment or may aggravate the effects of the drug.
* Subjects with systemic infection requiring antibiotics.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-10-28 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline body weight at week 8 | Week 0, Week 8
  Compared the difference of body weight between the week 8 and 0.

SECONDARY OUTCOMES:
Change from baseline body fat at week 8 | Week 0, Week 8
  Compared the difference of body fat between the week 8 and 0.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Jou Chien, PhD student, Principal Investigator — Chung Shan Medical University; Ying-Ching Feng, MS student, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, South, Taiwan